CLINICAL TRIAL: NCT01797354
Title: Impact of a Group Intervention on Breast Cancer Patient's Adjustment and Emotion Regulation at the End of Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: Jules Bordet Institute (Other)
Responsible Party: Principal Investigator, Prof. Isabelle Merckaert, PhD, professor, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Groupe support 22-007
Record Dates: First submitted 2011-12-28; First posted 2013-02-22 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: patients at the end of treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Cognitive Behavioral Therapy; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-behavioral therapy and hypnosis group (Experimental): Patients will receive (in groups of 6) fifteen 120-min sessions of group therapy including cognitive-behavioral techniques and hypnosis.
  Interventions: Behavioral: Cognitive-behavioral therapy and hypnosis group
- Support group (Active Comparator): Patients will receive (in groups of 6) fifteen 120-min support group session.
  Interventions: Behavioral: Support group

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy and hypnosis group
  Arms: Cognitive-behavioral therapy and hypnosis group
Behavioral: Support group
  Arms: Support group

SUMMARY:
Background: The end of treatment is for cancer patients the beginning of a critical rehabilitation period including numerous physical, emotional, professional and cognitive challenges. Specific interventions adapted to this post-treatment period need thus to be designed. Interventions such as group cognitive-behavioral therapy and hypnosis have been shown to be effective. However, moderate effect sizes, no comprehensive description of the treatment interventions and assessments relying only on self-report measures warrant further investigation. This study aims to assess, in breast cancer patients at the end of treatment, the impact of a group intervention combining cognitive-behavioral therapy and hypnosis versus a group intervention on patient's adjustment and emotion self-regulation.

Design: This is a two-armed, longitudinal, randomized controlled trial. Breast cancer patients finishing their radiation therapy treatment will be randomized to either an immediate group intervention combining cognitive-behavioral therapy and hypnosis or a group intervention. Patients will be assessed at three time points during the first year following the end of treatment: at 1 (T1), 6 (T2) and 12 (T3) months after the end of treatment. Patients' adjustment will be assessed through questionnaires. Patient emotion self-regulation ability will be assessed through their ability to respond both subjectively (self-reported emotional state) and objectively (heart rate) to two emotion self-regulation tasks.

Discussion: It is hypothesized that a group intervention combining cognitive-behavioral therapy and hypnosis will be more effective than a group intervention. Results of this study will contribute to improving post-treatment care for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic breast cancer (in situ or invesive)
* End of active treatments (surgery, chemotherapy and radiotherapy)
* No recurrence nor palliative care
* Min. 18 years
* Able to speak French
* Willing to be randomized to study intervention group
* Accept to give their written informed consent

Exclusion Criteria:

* No cognitive dysfunction
* No severe or uncontrolled psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Physical wellbeing: emotion regulation ability (heart rate, relaxation, quality of life,...) | Change from baseline in heart rate and relaxation ability at 6 (T2) and 12 months (T3)
  Questionnaires:
  * Quality of life questionnaires: "EORTC QLQ-C30" and "EORTC-BR23"
  * Edmonton symptom evaluation scale
  * Way of life questionnaire
Psychological wellbeing: emotional state, emotional adjustment, social adjustment, quality of life,... | Change from baseline in emotional state, emotional adjustment, social adjustment and quality of life at 6 (T1) and 12 (T2) months.
  Questionnaires:
  * the Hospital Anxiety and Depression Scale
  * the Rosenberg's Self-Esteem
  * the Mental Adjustment to Cancer Scale
  * the Fear of Cancer Recurrence Inventory
  * the Perceived Social Support Questionnaire
  * the Courtauld Emotional Control scale
  * the Ways of Coping Checklist
  * the Toronto Alexithymia Scale
  * a questionnaire about usual emotional state
  * a questionnaire about the use of relaxation techniques and self-hypnosis

CONTACTS AND LOCATIONS:
Overall Officials: Darius Razavi, Prof, Principal Investigator — Université Libre de Bruxelles, Institut Jules Bordet; Isabelle Merckaert, Prof, Principal Investigator — Université Libre de Bruxelles, Institut Jules Bordet
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

REFERENCES:
- [Derived] Merckaert I, Lewis F, Delevallez F, Herman S, Caillier M, Delvaux N, Libert Y, Lienard A, Nogaret JM, Ogez D, Scalliet P, Slachmuylder JL, Van Houtte P, Razavi D. Improving anxiety regulation in patients with breast cancer at the beginning of the survivorship period: a randomized clinical trial comparing the benefits of single-component and multiple-component group interventions. Psychooncology. 2017 Aug;26(8):1147-1154. doi: 10.1002/pon.4294. Epub 2016 Nov 7. PMID 27718533